CLINICAL TRIAL: NCT00898937
Title: Pilot Study for Analysis of Tumor Gene Expression by DNA Microarray Analysis in Patients Undergoing Breast Cancer Surgery or Core Biopsy Sampling
Brief Title: Gene Expression in Tumor Tissue From Women Undergoing Surgery for Breast Cancer or Core Biopsy of the Breast
Status: Terminated | Type: Observational
Why Stopped: Funding ended
Sponsor: Georgetown University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000377341; P50CA058185 (NIH); P30CA051008 (NIH); GUMC-99225
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Results first posted 2018-04-13 (Actual); Last update posted 2018-04-13 (Actual); Status verified 2018-02

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Microarray Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: microarray analysis — tumor specimen will be assessed by microarray analysis
Procedure: breast biopsy — A breast biopsy will be done to obtain a tumor specimen

SUMMARY:
RATIONALE: Studying samples of breast tissue in the laboratory may help doctors learn more about the genes and proteins found in breast tissue.

PURPOSE: This phase I trial is studying genes and proteins in breast tissue from women undergoing surgery for breast cancer or core biopsy of the breast.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess tumor gene expression information from women undergoing surgery for breast cancer or core biopsy sampling of the breast.

OUTLINE: This is a pilot study.

Tumor tissue is collected and analyzed for tumor gene expression by DNA microarray analysis for research studies.

PROJECTED ACCRUAL: A total of 100 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Undergoing surgery for breast cancer OR core biopsy sampling of the breast

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any woman undergoing a breast biopsy or breast surgery
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 1999-09; Primary Completion 2014-12 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claudine Isaacs, MD, Principal Investigator — Lombardi Comprehensive Cancer Center
Locations (1):
- Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Snap-frozen: Method of RNA recovery: Snap-frozen
  For more information about snap-frozen RNA recovery please see this link:
  https://www.thermofisher.com/us/en/home/references/ambion-tech-support/rna-isolation/tech-notes/effect-of-freeze-thawing-of-tissue-on-rna-integrity.html
- RNALater: Method of RNA recovery: RNALater
  For more information on RNAlater please see this link: https://www.thermofisher.com/us/en/home/brands/product-brand/rnalater.html
- FG002: Method of RNA recovery: unknown
Period: Overall Study
Arm/Group | Snap-frozen | RNALater | FG002
Started | 25 | 21 | 9
Completed | 25 | 21 | 9
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Snap-frozen: Method of RNA recovery: Snap-frozen
- RNALater: Method of RNA recovery: RNALater
- Unknown: Method of RNA recovery: unknown
- Total: Total of all reporting groups
Arm/Group | Snap-frozen | RNALater | Unknown | Total
Number analyzed (Participants) | 25 | 21 | 9 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 25 | 21 | 9 | 55
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 21 | 9 | 55
  Male | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Tumor Gene Expression as Assessed by RNA Microarray Analysis
Description: Concentration of RNA recovered from breast needle biopsies
Time Frame: 1 day
Measure: Mean (Standard Error); unit: micrograms
Arm/Group | Snap-frozen | RNALater | Unknown
Number analyzed (Participants) | 25 | 21 | 9
micrograms | 2.04 (0.51) | 3.49 (0.78) | 3.63 (0.48)

ADVERSE EVENTS:
Description: Serious and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Groups:
- EG002: Method of RNA recovery: unknown
Arm/Group | Snap-frozen | RNALater | EG002
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes